CLINICAL TRIAL: NCT04182399
Title: Role of Zonisamide in Advanced Parkinson's Disease (PD) in Egyptian Population: Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ali Shalash, professor of Neurology, Ain Shams University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MD282/2019
Record Dates: First submitted 2019-11-24; First posted 2019-12-02 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease, zonisamide, motor, fluctuation
MeSH Terms: conditions — Parkinson Disease | interventions — Zonisamide

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned to one of three groups: placebo group , ZNS group 25 mg and ZNS group 50 mg (30 patients each).In ZNS 50 mg group, ZNS will be started with a dose of 25 mg daily for one week then increased to 50 mg once daily to minimize side effects. Randomization was done by a research randomization program (https://www.randomizer.org), The copy of the randomization table of patients to the 3 groups was kept with 2 different personnel not working on the study.
  Amid to COVID19 and less access to patients in an advanced stage, a crossover design will be included SO patients in:
  Placebo arm will be randomized to arm 25 mg or 50 mg with at least 1-month washout Arm 25 mg & arm 50 mg will be shifted to placebo with at least 1 month washout
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: the PD will be randomized to 3 arms. Randomization was done by a research randomization, The copy of the randomization table of patients to the 3 groups was kept with 2 different personnel not working on the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients 25 ZNS (Active Comparator): 30 patients receive oral 25 mg ZNS daily
  Interventions: Drug: Zonisamide Capsules
- Patients 50 ZNS (Active Comparator): 30 patients receive oral 50 mg ZNS daily
  Interventions: Drug: Zonisamide Capsules
- Patients Placebo (Placebo Comparator): 30 patients receive placebo
  Interventions: Drug: Zonisamide Capsules

INTERVENTIONS:
Drug: Zonisamide Capsules — anti-epileptic drug that recently used as add on therapy of wearing off and fluctuation complications of dopaminergic drugs in PD patients
  Other Names: Convagran

SUMMARY:
Zonisamide (ZNS) (1,2-Benzisoxazole-3-methanesulfonamide) is an anti-epileptic drug. In three double blinded placebo controlled studies, ZNS- as an adjunctive treatment- showed beneficial effects on motor symptoms of PD with a low incidence of adverse events. As a result 25 mg daily of ZNS was approved in 2009 in Japan as an adjunctive treatment in PD patients whose condition responded insufficiently to Levodopa treatment.

Most observations of a beneficial effect of ZNS have been in Japanese people, and the antiparkinsonian mechanism of action is unclear. So, ZNS is a promising but still investigational drug to treat PD and more studies are warranted.

this study will investigate the efficacy and tolerability of Zonisamide as an adjunctive treatment in Egyptian patients with advanced PD, including motor fluctuations, levodopa induced dyskinesia and existing nonmotor symptoms. Additionally it investigates its effects on quality of life of PD patients.

DETAILED DESCRIPTION:
Type of Study: Randomized double blinded Placebo controlled study.

* Study Setting: Movement disorders clinic of neurology department, Ain Shams University Hospitals.
* Study Period : 2 years.
* Study Population: Patients with advanced PD and insufficient response to dopaminergic drugs .

Inclusion Criteria:

* Age older than 18 years of both male and female genders.
* Individuals diagnosed with PD based on the presence of 2 of 3 cardinal features & United Kingdom bank criteria for idiopathic Parkinson's disease.
* Patients with manifestations of advanced PD defined according to the consensus on the definition of advanced PD.
* Inadequate response to dopaminergic medications due to limitations related to side effects, or levodopa related long-term problems as wearing-off phenomena, "on"-"off" fluctuation, levodopa induced dyskinesia and freezing phenomena, no-"on" and delayed-"on,".

Exclusion Criteria:

1. Patients with atypical or secondary parkinsonian syndromes excluding PD.
2. Patients who could not perform the tests.
3. Women who were or might be pregnant, who did not practice effective contraception and were of childbearing potential, or who were breastfeeding.

Ethical Considerations:

All of the patients will be informed of the objectives, procedures and possible benefits and risks of the study and will provide written voluntary consent.

The study will conform to the standards of the Ethical Review Committee, Ain Shams University.

Study Procedures:

- Patients diagnosed with PD will be evaluated for inclusion and exclusion criteria. Eligible patients will be randomly assigned to one of three groups: placebo group , ZNS group 25 mg and ZNS group 50 mg (30 patients each).In ZNS 50 mg group, ZNS will be started with a dose of 25 mg daily for one week then increased to 50 mg once daily to minimize side effects. The dosage and regimen of ongoing antiparkinsonian drugs and other drugs that may affect PD symptoms will remain unchanged one month before and through the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1 -Age older than 18 years of both male and female genders. 2-Individuals diagnosed with PD based on the presence of 2 of 3 cardinal features & UK bank criteria for idiopathic Parkinson's disease. 3-Patients with motor complications of PD (Hoehn and Yahr stage 2-3)(on therapy) and at least 2 hours off time.

Exclusion Criteria:

1 -Patients with atypical or secondary Parkinsonism syndromes excluding PD. 2-Patients who could not perform the tests. 3-Women who were or might be pregnant, who did not practice effective contraception and were of childbearing potential, or who were breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Off motor daily time | at 1 and 3 months
  assessing change of Off and on time using Movement Disorders Society- Unified Parkinson's Disease Rating Scale (MDS UPDRS)
levodopa related Dyskinesia | at 1 and 3 months
  Dyskinesia will also be evaluated with Movement Disorders Society- Unified Dyskinesia Rating Scale (MDS-UDysRS)

SECONDARY OUTCOMES:
Quality of life (daily life activities) | at 3 months
  parkinson disease questionnaire-39
cognitive outcome | at 3 months
  using Montreal cognitive assessment
The non-motor symptoms scales | at 1 and 3 months
  using The non-motor symptoms scales (NMSS)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Shalash, PhD, Principal Investigator — Department of Neurology, Faculty of Medicine, Ain Shams Univeristy
Locations (2):
- Egypt (2):
  - Department of Neurology, Ain Shams University Hospital, Cairo, Abbasia
  - Ain Shams Univeristy, Cairo

REFERENCES:
- [Derived] Essam M, Hamid E, Abushady E, El-Balkimy M, Antonini A, Shalash A. Role of zonisamide in advanced Parkinson's disease: a randomized placebo-controlled study. Neurol Sci. 2024 Apr;45(4):1725-1734. doi: 10.1007/s10072-024-07396-w. Epub 2024 Feb 20. PMID 38376645